CLINICAL TRIAL: NCT04329572
Title: Open, Multicentric, Non Randomized, Exploratory Clinical Trial to Assess the Efficacy and Safety of Hydroxychloroquine and Azithromycin for the Treatment of Acute Respiratory Syndrome (COVID-19) Caused by SARS-CoV-2 Virus
Brief Title: Efficacy and Safety of Hydroxychloroquine and Azithromycin for Patients With Moderate to Severe COVID-19
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Azidus, the CRO hired for this study by Prevent Senior has lost the interest to conduct this study.
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIAPRE0320OR
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: All patients included in the study will receive hydroxychloroquine (HCQ) 400 mg (BID/ 7 days) and azithromycin (AZT) (500 mg/ 5 days) on top of standard care. Patients that do not consent to participate or that do not fulfill eligibility criteria will be invited to participate as control group and will receive standard care only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCQ + AZT (Experimental): All patients included in the study will receive HCQ (400 mg BID on D1 and 400 mg/day on D2 to D5) and AZT (500 mg/ 5 days) on top of standard care.
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Azithromycin Tablets

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — All patients included in the study will receive HCQ (400 mg BID on D1 and 400 mg/day on D2 to D5) for 5 days.
  Other Names: Reuquinol
Drug: Azithromycin Tablets — All patients included in the study will receive AZT 500 mg per day for 5 days.
  Other Names: Azithromycin

SUMMARY:
This is an exploratory study to evaluate the efficacy of hydroxychloroquine (400 mg BID on D1 and 400 mg/day on D2 to D5) and azithromycin (500 mg/ 5 days) to treat moderate to severe COVID-19 pneumonia.

DETAILED DESCRIPTION:
This is an exploratory, open label, multi-center study to evaluate the efficacy of hydroxychloroquine (HCQ) (400 mg BID on D1 and 400 mg/day on D2 to D5) and azithromycin (AZT) (500 mg/ 5 days) to treat moderate to severe COVID-19 pneumonia.

We aim to demonstrate decrease in hospital related complications among patients who are hospitalized with moderate or severe COVID-19 by treating them with HCQ and AZT on top of standard care compared to patients who receive standard care only.

Patients hospitalized with confirmed diagnosis of COVID-19 will receive the treatment.

Patients that do not fulfill the inclusion/exclusion criteria or that is not willing to participate in the study will be invited to consent the use of their data as part of a "control" group.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from patient or legal representative.
2. Male or female, aged ≥ 18 years;
3. Laboratory confirmation of 2019-nCoV infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source;
4. At least one of the characteristic symptoms of COVID-19
5. Hospitalized for up to 36h with non-invasive ventilation or up to 24h with invasive ventilation.
6. Negative result for pregnancy test (if applicable).

Exclusion Criteria:

1. Participating in another RCT in the past 12 months;
2. Known allergy to HCQ or chloroquine
3. Any contraindication to HTC or AZT, including retinopathy and prolonged QT,
4. Severely reduced LV function
5. Severely reduced renal function;
6. Pregnancy or breast feeding
7. Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of the investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of acute respiratory syndrome, oxygen saturation hemodynamic stability | 28 days
  Evaluation of change from baseline. Kaplan-meier method will be used.

SECONDARY OUTCOMES:
Viral load | Day 6
  Evaluation of change in viral load
Change in Clinical Condition | 28 days
  Time for normalization of body temperature, respiratory rate and cough relief
Evolution of Acute Respiratory Syndrome | 28 days
  Time to wean off oxygen supplementation and / or invasive / non-invasive ventilatory support;
Hospital discharge | 28 days
  Time to be discharged from hospital
Rate of mortality within 28-days | 28 days
  Evaluation of change in acute respiratory syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Ferrara, Study Director — Azidus Brasil
Locations (1):
- Prevent Senior Private Operadora de Saúde LTDA., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.